CLINICAL TRIAL: NCT02361723
Title: A Phase 1A/1B, Open Label, Multiple Dose, Dose Escalation, and Expansion Study to Investigate the Safety, Pharmacokinetics, Food Effect, and Antitumor Activities of BGB-290 in Subjects With Advanced Solid Tumors
Brief Title: Phase 1a/1b BGB-290 for Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-290-AU-002
Record Dates: First submitted 2015-01-29; First posted 2015-02-12 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: For Participants With Advanced Solid Tumors Failed With Previous Lines of Treatment
Keywords: Advanced Solid Tumors
MeSH Terms: interventions — pamiparib

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (5):
- ovarian cancer, fallopian cancer, or primary peritoneal cancer (Experimental): 60mg BID oral.
  Interventions: Drug: BGB-290
- Breast Cancer (Experimental): 60mg BID Ora
  Interventions: Drug: BGB-290
- Prostate Cancer (Experimental): 60mg BID Oral
  Interventions: Drug: BGB-290
- Small Cell Lung Cancer (Experimental): 60mg BID Oral
  Interventions: Drug: BGB-290
- Gastric Cancer (Experimental): 60mg BID Oral
  Interventions: Drug: BGB-290

INTERVENTIONS:
Drug: BGB-290
  Arms: ovarian cancer, fallopian cancer, or primary peritoneal cancer
Drug: BGB-290
  Arms: Breast Cancer
Drug: BGB-290
  Arms: Prostate Cancer
Drug: BGB-290
  Arms: Small Cell Lung Cancer
Drug: BGB-290
  Arms: Gastric Cancer

SUMMARY:
The study contains Phase 1A and Phase 1B. Phase 1A has Part1 (BID Dose Escalation) and Part2 (QD Dosing Escalation) Evaluation of a cohort of at least three participants completing one cycle of treatment at that dose level and dose regimen is required prior to determining the next dose level and dose regimen for the next cohort. Phase 1B has PartA (BID Dosing Expansion) will investigate efficacy in participants with selected tumor types and further evaluate safety and tolerability of BGB 290 at recommended dose for future studies. and PartB (Food Effect) will investigate the food effect on the Pharmacokinetics (PK) of BGB 290 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study contains Phase 1A and Phase 1B. Phase 1A has Part1 (BID Dose Escalation) and Part2 (QD Dosing Escalation) Evaluation of a cohort of at least three participants completing one cycle of treatment at that dose level and dose regimen is required prior to determining the next dose level and dose regimen for the next cohort. Phase 1B has PartA (BID Dosing Expansion) will investigate efficacy in participants with selected tumor types and further evaluate safety and tolerability of BGB 290 at recommended dose for future studies. and PartB (Food Effect) will investigate the food effect on the PK of BGB 290 in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female and at least 18 years of age with a life expectancy of at least 12 weeks.
2. Histologically or cytologically confirmed malignancy that has progressed to the advanced or metastatic stage for which no effective standard therapy is available.
3. BRCA1/2 mutations are not required but enrichment of this participant population is permitted.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
5. Adequate bone marrow, liver, and renal function.
6. Participants who have histologic or cytologic confirmation of malignancy that has progressed to the advanced or metastatic stage.
7. Eligible participants who have received the prior chemotherapy regimen in the advanced or metastatic setting.
8. Females of childbearing potential unwilling to use a highly effective method of contraception during treatment and throughout the study until 28 days after the last investigational product administration.
9. Able to swallow and retain oral medication.

Key Exclusion Criteria:

1. Participants did not receive prior therapies targeting poly-ADP ribose polymerase (PARP).
2. Participants who are not considered to be refractory to platinum-based therapy (e.g., progressive disease at the first tumor assessment while receiving platinum treatment).
3. Participants who have not been treated with chemotherapy, biologic therapy, immunotherapy, or other investigational agent within five times half-lives of the last treatment or within 4 weeks (whichever is longer) prior to starting study drug (or who have not recovered from the side effects of such therapy).
4. Participants who have not undergone major surgery/surgical therapy for any cause within 4 weeks of screening visit.
5. Participants must have recovered from the treatment and have a stable clinical condition before entering this study.
6. Participants who have not received therapeutic radiotherapy to target lesions. 7.Participants who have received local palliative radiotherapy of non-target lesions for local symptom control within the last 21 days must have recovered from any adverse effects of radiotherapy before recording screening symptoms. 8.No untreated brain metastasis or unstable neurologic condition after the completion of radiation, or requiring corticosteroid of > 40 mg prednisone daily equivalent dose to control the symptoms.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate ([ORR]: Complete Response (CR) + Partial Response (PR)) based on RECIST Version 1.1 | through study completion, an average of 1 year
  The primary endpoint of the study was a composite response rate that included ORR, a ≥50% decrease in serum prostate-specific antigen (PSA), and/or a decrease in circulating tumor cells.
Prostate-specific antigen (PSA) response (for prostate cancer participants only) based on Prostate Cancer Working Group 2 (PCWG2) criteria | through study completion, an average of 1 year
  The primary endpoint of the study was a composite response rate that included ORR, a ≥50% decrease in serum prostate-specific antigen (PSA), and/or a decrease in circulating tumor cells.
Primary PK 1 | through study completion, an average of 1 year
  Primary PK parameter is area under the plasma concentration time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUClast).
Primary PK 2 | through study completion, an average of 1 year
  Primary PK parameter is area under plasma concentration time curve (AUC).
Primary PK 3 | through study completion, an average of 1 year
  Primary PK parameter is maximum observed plasma concentration (Cmax).

SECONDARY OUTCOMES:
Progression free survival | through study completion, an average of 1 year
  Participants, who are withdrawn from the study without documented progression, will be censored at the date of the last tumor assessment when the participant was known to be progression free. Participants without post screening tumor assessments, but known to be alive will be censored at the time of the first administration of BGB 290).
Duration of response for responders (CR or PR) and duration of SD (defined only for participants whose confirmed best response is CR, PR, or SD. | through study completion, an average of 1 year
  For participants who are alive without progression following the qualifying response, duration of response will be censored on the date of last evaluable tumor assessment or last follow up for progression of disease).
The number and proportion of participants who achieve objective tumor response (complete response [CR], partial response [PR], and CR+PR) or stable disease (SD). | through study completion, an average of 1 year
  For ovarian cancer participants, tumor responses may also be evaluated using RECIST Version 1.1 combined with CA-125 based on the Gynecologic Cancer Intergroup (GCIG) criteria. For participants with prostate cancer, PCWG2 criteria may be used to evaluate responses by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millward, MD, Principal Investigator — Linear Clinical Research
Locations (7):
- Australia (7):
  - Gosford Hospital, Gosford, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Flinders Medical Centre, Bedford PK, South Australia
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lickliter JD, Gan HK, Meniawy T, Yang J, Wang L, Luo LS, Millward M. A phase I dose-escalation study of BGB-290, a novel PARP1/2 selective inhibitor in patients with advanced solid tumors. Journal of Clinical Oncology. 2016; 34(15): DOI: 10.1200/JCO.2016.34.15_suppl.e17049
- [Derived] Lickliter JD, Voskoboynik M, Mileshkin L, Gan HK, Kichenadasse G, Zhang K, Zhang M, Tang Z, Millward M. Phase 1A/1B dose-escalation and -expansion study to evaluate the safety, pharmacokinetics, food effects and antitumor activity of pamiparib in advanced solid tumours. Br J Cancer. 2022 Mar;126(4):576-585. doi: 10.1038/s41416-021-01632-2. Epub 2021 Nov 18. PMID 34795408
- [Derived] Xu B, Yin Y, Dong M, Song Y, Li W, Huang X, Wang T, He J, Mu X, Li L, Mu S, Zhang W, Li M. Pamiparib dose escalation in Chinese patients with non-mucinous high-grade ovarian cancer or advanced triple-negative breast cancer. Cancer Med. 2021 Jan;10(1):109-118. doi: 10.1002/cam4.3575. Epub 2020 Oct 31. PMID 33128299